CLINICAL TRIAL: NCT04858984
Title: Virtual Reality, Experience During Labour; a Qualitative Research
Brief Title: Virtual Reality, Experience During Labour; a Qualitative Research (VIREL)
Acronym: VIREL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, Anne-Claire Musters, Principal Investigator, Zuyderland Medisch Centrum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL-METCZ20200096
Record Dates: First submitted 2021-04-11; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Labor Pain; Virtual Reality; Analgesia; Pain
Keywords: Virtual reality; labour pain; analgesia; obstetric care
MeSH Terms: conditions — Labor Pain; Agnosia; Pain

STUDY DESIGN:
Intervention Model Description: Qualitative research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality group (Experimental): All participants experienced an immersive guided meditation virtual reality (VR1) and an interactive game virtual reality (VR2) experience during labour. Both VR interventions were offered for 10 minutes. Before and immediately after an intervention, the patient was asked to fill out a Numeric Rating Scale (NRS) score for pain.
  During the 30-minute intermission after the VR intervention the patient completed the post-intervention questionnaire.
  VR1 consisted of a video of an exotic location guided by the sound of the waves and a calm English-speaking voice. VR2 required women to use the controller to throw snowballs in order to catch presents and reach the next level. Patients were allowed to stop using the VR at any moment during the intervention.
  Five days post-partum all participants who completed both VR interventions were contacted by telephone for an interview.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — A portable, standalone VR headset called Oculus Go (Facebook Technologies, LLC. 1601 Willow Road, Menlo Park, CA 940250) with a head-mounted display with built in audio drivers was used. Disposable hygiene masks and a surgical cap were used as an underlay below the headset an

SUMMARY:
Childbirth is associated with labour pain and can be regarded as one of the most serious kinds of pain. Labour pain management methods include pharmacological and non-pharmacological methods. There is increasing evidence that virtual reality (VR) is effective in the reduction of labour pain.

The aim of this qualitative study is to explore the experience, preference, and satisfaction of the use of two different VR scenario's during labour. The secondary outcome parameter is the effect of VR on pain reduction and anxiety during labour, measured by NRS score.

DETAILED DESCRIPTION:
Epidural Analgesia (EA) has been regarded as the most effective method of labour analgesia. Pharmacological analgesia methods are known to have adverse side effects, such as nausea, vomiting and drowsiness in parental opioids; pruritus, nausea, desaturation, respiratory depression and apnea in patient-controlled remifentanil analgesia; and maternal fever, maternal hypotension and urinary retention in EA. Furthermore, routine EA is likely resulting in more operative deliveries. Considering these possible adverse effects, it is worth exploring alternative methods for labour pain relief.

There is increasing evidence that virtual reality (VR) is effective in the reduction of labour pain.

This VIREL study aims to examine the experience, preference, and satisfaction of VR in women during labour. The study is set up as a single centre, qualitative study in a non-university teaching hospital in The Netherlands with 2800 deliveries annually. Participants will experience an immersive guided relaxation VR (VR1) and an interactive game (VR2) during labour. VR1 consists of a video of an exotic location guided by the sound of the waves and a calm English-speaking voice. VR2 requires women to use the controller to throw snowballs in order to catch presents and reach the next level. Patients are allowed to stop using the VR at any moment during the intervention.

When the participant is declared to be in labour, defined as having regular painful uterine contractions, cervical effacement and at least 3cm dilatation, VR1 will be offered for ten minutes. Before and immediately after VR1, the patient is asked to fill out a Numeric Rating Scale (NRS) score for pain.

During the 30-minute intermission after VR1 the patient fills out the post-intervention questionnaire regarding VR1. Subsequently, VR2 is offered for ten minutes. Before and immediately after VR2 the patient filled in the NRS score for pain, and the patient completed a post-intervention questionnaire regarding VR2. Additional use of VR is allowed by maternal request. Five days post-partum all participants who completed both VR interventions will be contacted by telephone for a semi-structured interview.

ELIGIBILITY:
Inclusion Criteria:

* Written and orally given informed consent
* 18 years and older
* Native Dutch speaker
* Pregnant of a singleton in cephalic presentation
* Intention to deliver vaginally
* Induced labour by a balloon or artificial rupture of membranes

Exclusion Criteria:

* Chronic pain patients; defined as 'persistent or recurrent pain lasting longer than 3 months'. The pain is not due to the gynecological problem.
* Chronical use of pain medication (opioids)
* Alcohol or drug abuse
* Known car sickness or susceptibility to motion sickness
* Epileptic insults in previous history
* Psychotically seizures in previous history
* Claustrophobic
* Blindness
* History of mental illness
* Severe hearing or vision deficits
* Epidural Anesthesia during labour

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women.
Enrollment: 28 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Patients' VR experience, satisfaction and application preference regarding the guided meditation VR | During labour: directly after the first VR intervention (Guided meditation VR)
  A patients' VR experience, satisfaction and application preference was examined using a post-intervention questionnaire.
  A short post intervention questionnaire, intended to provide a first feedback about the experience and preference of the VR application the patient used a few minutes ago. Ratings varied of very pleasant (+5) versus very unpleasant (0) and very much (+5) versus not at all (0).
  Theme's: General experience of VR1 (meditation) / VR2 (game), the amount of distraction, feeling of anxiety during VR1 (meditation) / VR2 (game), reusing VR1 (meditation) / VR2 (game), preference of environment (beach environment or do you prefer something else?), side effects.
Patients' VR experience, satisfaction and application preference (meditation or interactive game) | 5 days after labour
  A patients' VR experience, satisfaction and application preference was examined using a semi-structured interview.
  Theme's of the semi-structured interview:
  1. VR experience
  * General experience
  * VR1 experience
  * VR2 experience
  * Side effects
  * Reusing VR
  * Recommendation to other women
  * Improvements
    2 Pain reduction
  * Pain intensity
  * Pain perception
  * Distraction
    3 Usability VR application
  * VR application
  * Comfort of VR glasses
Patients' VR experience, satisfaction and application preference regarding the interactive game | During labour: directly after the first VR intervention (Interactive game)
  A patients' VR experience, satisfaction and application preference was examined using a post-intervention questionnaire.
  A short post intervention questionnaire, intended to provide a first feedback about the experience and preference of the VR application the patient used a few minutes ago. Ratings varied of very pleasant (+5) versus very unpleasant (0) and very much (+5) versus not at all (0).
  Theme's: General experience of VR1 (meditation) / VR2 (game), the amount of distraction, feeling of anxiety during VR1 (meditation) / VR2 (game), reusing VR1 (meditation) / VR2 (game), preference of environment (beach environment or do you prefer something else?), side effects.

SECONDARY OUTCOMES:
Labour pain | 4 moments during labour: Before the first VR intervention (meditation), directly after the first VR intervention (meditation). Before the second VR intervention (game), directly after the second VR intervention (game).
  Labour pain before and directly after VR was evaluated using the Numeric (pain) rating scale (The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).)

CONTACTS AND LOCATIONS:
Overall Officials: Martine Wassen, M.D., Principal Investigator — Zuyderland MC
Locations (1):
- Zuyderland MC, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available at the moment. The study protocol, statistical analysis plan and informed consent form will be available after publication of the article.

REFERENCES:
- [Derived] Musters A, Vandevenne AS, Franx A, Wassen MMLH. Virtual Reality Experience during Labour (VIREL); a qualitative study. BMC Pregnancy Childbirth. 2023 Apr 24;23(1):283. doi: 10.1186/s12884-023-05432-9. PMID 37095433